CLINICAL TRIAL: NCT00927303
Title: Comparison of Quality and Reproducibility of Retinal Thickness Measurements in Two Spectral Domain OCT- Machines
Brief Title: The Spectralis-Cirrus Study
Status: Completed | Type: Observational
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Ilse Krebs, MD, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Other Study IDs: 09-086-0609
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Exudative Age Related Macular Degeneration
Keywords: retinal thickness; threshold algorithm; optical coherence tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — male or femal persons age over 50 years with exudative age-related macular degeneration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Group 1: Intervention 1 Sequence of observers: observer1, observer 2, observer 1, observer 2
  Interventions: Device: Cirrus-Spectralis
- group 2: intervention 1 sequence of observers: observer 2, observer 1, observer 2, observer 1
  Interventions: Device: Cirrus-Spectralis
- group 3: intervention 2 sequence of observers: 1,2,1,2
  Interventions: Device: Spectralis-Cirrus
- group 4: intervention 2 sequence of observers: 2,1,2,1
  Interventions: Device: Spectralis-Cirrus
- group 5: intervention 1 sequence of observers 1,1,2,2
  Interventions: Device: Cirrus-Spectralis
- group 6: intervention 1 sequence of observers 2,2,1,1
  Interventions: Device: Cirrus-Spectralis
- group 7: intervention 2 sequence of observers: 1,1,2,2
  Interventions: Device: Spectralis-Cirrus
- group 8: intervention 2 sequence of observers: 2,2,1,1
  Interventions: Device: Spectralis-Cirrus

INTERVENTIONS:
Device: Cirrus-Spectralis — 512x128 cúbe program of Cirrus OCT first retinal volume 121 line of Spectralis OCT thereafter
  Groups: Group 1; group 2; group 5; group 6
Device: Spectralis-Cirrus — retinal volume program 121 lines Spectralis OCT first 512x128 program Cirrus OCT thereafter
  Groups: group 3; group 4; group 7; group 8

SUMMARY:
Retinal thickness measurement is one of the most important examinations in the follow up of exudative age-related macular degeneration. Prior studies have shown that there are a series of algorithm line failures in OCT examinations. This study is conducted to compare the quality of the examinations of to different spectral domain OCT machines concerning the positioning of algorithm lines. Furthermore the reproducibility of the examinations id tested, both machines provide different techniques to guarantee that in repeated examinations the same location is examined.

ELIGIBILITY:
Inclusion Criteria:

* Exudative age related macular degeneration

Exclusion Criteria:

* Macular pathologies other than age related macular degeneration (diabetic maculopathy, macular pucker, macular hole,
* Visualization of the macula not possible (dens cataract, vitreous haemorrhage)
* Not consented patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female persons aged more than 50 years with exudative age related macular degeneration
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of examinations with correctly set threshold algorithm lines | 1 day

SECONDARY OUTCOMES:
Differences of mean retinal thickness in the central region | 1 day
Differences of retinal volume | 1 day
Distance acuity | 1 day
Age | 1 day
Classification of the lesion | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, MD, Prof, Study Chair — Ludwig Boltzmann Institute for Retinology and Biomicroscopic Laser Surgery
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Krebs I, Smretschnig E, Moussa S, Brannath W, Womastek I, Binder S. Quality and reproducibility of retinal thickness measurements in two spectral-domain optical coherence tomography machines. Invest Ophthalmol Vis Sci. 2011 Sep 1;52(9):6925-33. doi: 10.1167/iovs.10-6612. PMID 21791591